CLINICAL TRIAL: NCT03781934
Title: A Phase 1/2a Study in 3 Parts to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of MIV-818 in Patients With Liver Cancer Manifestations
Brief Title: A Study to Evaluate MIV-818 in Patients With Liver Cancer Manifestations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MIV-818-101/201
Record Dates: First submitted 2018-11-07; First posted 2018-12-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma; Liver Metastases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: Intrapatient dose escalations continuing into interpatient dose escalations to end with dose expansion cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIV-818 (fostroxacitabine bralpamide) + pembrolizumab (Experimental): Phase 2a expansion cohort HCC
  Interventions: Drug: MIV-818 (fostroxacitabine bralpamide) + pembrolizumab
- MIV-818 (fostroxacitabine bralpamide) + lenvatinib (Experimental): Phase 2a expansion cohort HCC
  Interventions: Drug: MIV-818 (fostroxacitabine bralpamide) + lenvatinib

INTERVENTIONS:
Drug: MIV-818 (fostroxacitabine bralpamide) + pembrolizumab — MIV-818 - oral capsules; pembrolizumab - IV
  Arms: MIV-818 (fostroxacitabine bralpamide) + pembrolizumab
Drug: MIV-818 (fostroxacitabine bralpamide) + lenvatinib — MIV-818 - oral capsules; lenvatinib - oral capsules
  Arms: MIV-818 (fostroxacitabine bralpamide) + lenvatinib

SUMMARY:
This is an open-label, multicentre dose escalation/expansion study to assess safety and tolerability of MIV 818 as either monotherapy or in combination with 1) lenvatinib, a tyrosine kinase inhibitor used as a standard of care for the treatment of HCC or 2) pembrolizumab, a PD-1 inhibitor. The monotherapy parts of the study will include patients with various solid tumours that have spread to the liver, or alternatively originating in the liver. Evaluations of MIV-818 in combination with lenvatinib or pembrolizumab will only include patients with HCC.

DETAILED DESCRIPTION:
This study will be conducted in three phases. The initial phase, 1a, will enroll up to 12 subjects and include a total of one dose escalation per patient. Once pre-defined criteria for starting phase 1b monotherapy has been met among the enrolled patients in phase 1a, the next phase of the study will be initiated. Phase 1b monotherapy will enroll up to 30 patients in a 3+3 design with interpatient dose escalations. All dose escalation decisions will be made by a safety review committee that will meet regularly during the study conduct. When the MTD has been established, the SRC will provide a RP2D for monotherapy. Phase 1b combination constitutes an interpatient dose escalation to identify the RP2D for MIV-818 when used in combination with 1) lenvatinib and 2) pembrolizumab therapy. This part of the study will enroll up to 36 patients in a 3+3 design with interpatient dose escalations. Safety review will be performed by the SRC to determine the RP2D of MIV 818 for use in combination with lenvatinib and pembrolizumab. The SRC may recommend that the selected dose of MIV-818 is further evaluated in up to 30 patients in the Phase 2a expansion part of the study.

ELIGIBILITY:
Inclusion criteria:

1. Male or female ≥ 18 years of age on the day of signing informed consent.
2. Able to understand and voluntarily sign a written informed consent and is willing, and able, to comply with the protocol requirements.
3. Must have measurable disease based on RECIST v1.1 as determined by the site study team. Must have at least 1 target lesion in the liver. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
4. Must have a Child-Pugh A status for Phase 1a and a Child-Pugh A or B status for Phase 1b and 2a. SRC discretion to restrict to Child-Pugh A status for Phase 1b and 2a.
5. Must have an ECOG performance status of 0 or 1 at Screening.
6. Must have life expectancy of > 12 weeks in the investigator's opinion.
7. Must have ALT and AST ≤ 5.0 × upper limit of normal (ULN) at Screening.
8. Must have total bilirubin (TBil) ≤ 3.0 mg/dL at Screening.
9. Must have adequate renal function with estimated creatinine clearance

   ≥ 60 mL/min (based on Cockcroft and Gault formula or similar) at Screening
10. Must have platelets ≥ 75,000/mL at Screening.
11. Must have International Normalized Ratio (INR) ≤ 1.7 at Screening. Female who is postmenopausal, OR Female who is of childbearing potential (postmenarchal) who agrees to use a highly efficient method of contraception (ie, a method with less than 1% failure rate [eg, sterilization, hormone implants, hormone injections, intrauterine devices, or vasectomized partner or combined birth control pills]) from Screening until 90 days after the final dose of MIV-818.

OR Male who agrees to use condoms from Screening until 90 days after the final dose of MIV-818.

OR Male with a female partner of childbearing potential (WOCBP) who is using a highly efficient method of contraception as described above.

13. WOCBP must have a negative serum pregnancy test at Screening and negative (serum or urine) pregnancy test within 72 h before the first study drug dose.

Phase 1a and 1b specific Inclusion Criteria:

14. Must have progressed on or are intolerant of standard therapy with:

1. Histologically or cytologically confirmed HCC, including fibrolamellar HCC; patients with HCC that received their diagnosis according to the agreed international radiological guideline are also admissible upon agreement between the investigator and the medical monitor, or
2. Histologically or cytologically confirmed iCCA, or
3. Liver metastases from colon, rectal, or gastric solid tumors with limited extrahepatic tumor burden (any extrahepatic metastases should be limited to 1 other site and a maximum of 1 target lesion outside the liver).

Phase 1b Monotherapy-specific Inclusion Criterion:

15. Must have:

1. Histologically or cytologically confirmed HCC, including fibrolamellar HCC; patients with HCC that received their diagnosis according to the agreed international radiological guideline are also admissible upon agreement between the investigator and the medical monitor, or
2. Histologically or cytologically confirmed iCCA, or
3. Liver metastases from solid tumors, with limited extrahepatic tumor burden (i.e. no brain or bone metastases), any extrahepatic metastases should be limited to 1 other site and a maximum of 1 target lesion outside the liver).

   Combination therapy-specific Inclusion Criterion:

   16. Must have histologically or cytologically confirmed HCC that is considered advanced or unresectable, i.e. not suitable for either surgery, radiofrequency ablation (RFA) or loco-regional therapies (patients with HCC that received their diagnosis according to the agreed international radiological guideline are also admissible upon agreement between the investigator and medical monitor). Patients with fibrolamellar HCC or a mixed HCC and iCCA will be excluded.

   17. Must have progressed on or are intolerant of 1or 2 lines of standard therapy for HCC (see also exclusion criterion no. 20) and are now candidates for lenvatinib or pembrolizumab treatment.

   Exclusion Criteria:
   1. Tumor volume exceeding 50% of liver.
   2. History of previous malignancy within the last 5 years except basal cell carcinoma or carcinoma in situ in solid organ.
   3. Known CNS or brain metastases, unless previously treated and stable for 3 months.
   4. Ongoing significant disease other than target disease as judged by the investigator to compromise the patients' ability to complete this study.
   5. History of solid organ transplant or bone marrow transplant.
   6. Receiving immunosuppressive therapy including oral corticosteroids.
   7. Active hepatitis B (eg, hepatitis B surface antigen [HBsAg] reactive) and patients with active hepatitis C (eg, hepatitis C RNA is [qualitative] detected).
   8. Positive human immunodeficiency virus (HIV) infection.
   9. Poorly controlled ascites and/or requirement for therapeutic paracentesis more frequently than once every 3 months.
   10. Symptomatic encephalopathy within 3 months prior to Screening and/or requirement for medication for encephalopathy.
   11. Esophageal variceal bleeding within 2 weeks prior to Screening.
   12. Receiving prior anticancer therapy within 4 weeks prior to first dose of MIV-818.
   13. Receiving any other investigational agent within 4 weeks prior to Screening
   14. Enrolled in another clinical study with an investigational drug.
   15. Presence of residual toxicities of CTCAE Grade > 1 after prior anticancer therapy within 2 weeks of first treatment with MIV-818, except for alopecia.
   16. History of allergic reactions attributed to compounds of similar chemical or biological composition to MIV-818.
   17. HCC of diffuse infiltrative type.
   18. Receiving drugs that are extensively metabolized by cytochrome P450 (CYP) 3A4 that have a narrow therapeutic index. Drugs that are extensively metabolized by CYP3A4 that have a narrow therapeutic index must be discontinued 5 half-lives before first dose of MIV-818.

       Combination therapy-specific Exclusion Criteria:

       Patients are excluded from combination therapy parts of this study if any of the following criteria are met:
   19. Patients with a diagnosis of fibrolamellar HCC.
   20. Received >2 lines of therapy for the treatment of advanced HCC.
   21. Systolic blood pressure (BP) ≥160 mmHg or diastolic BP ≥100 mmHg despite optimal anti-hypertensive therapy and with no change in anti hypertensive agents within the last 1 week prior to Screening.
   22. Women who are breastfeeding.
   23. Bleeding disorders or receiving anti-coagulation drugs.
   24. Any interventional treatment for esophageal varices required within 28 days of study treatment.
   25. Hepatic encephalopathy in the last 6 months.
   26. QTc interval is greater than 480 milliseconds at Screening.
   27. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
   28. Has an active infection requiring systemic therapy.

       Exclusion criteria applicable to pembrolizumab cohort only:
   29. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to planned start of study therapy.
   30. Presence of known active tuberculosis (TB; Bacillus tuberculosis).
   31. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
   32. Known history of, or any evidence of active, non-infectious pneumonitis or has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.

       Exclusion criterion applicable to lenvatinib cohort only:
   33. Proteinuria > 1g / 24 hours. Patients with > 1+ proteinuria on dipstick testing will need a 24-hour urine protein measured to exclude proteinuria > 1g / 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Percentage of participants with an adverse event, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0
Incidence and magnitude of clinically significant changes in red blood cell count, white blood cell count and platelet count | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Change from baseline
Incidence and magnitude of clinically significant changes in aspartate aminotransferase (AST) and alanine aminotransferase (ALT) | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Change from baseline
Incidence and magnitude of clinically significant changes in bilirubin | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Change from baseline
Incidence of clinically significant changes in vital sign - Systolic and diastolic blood pressure | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Millimeter of mercury (mmHg)
Incidence of clinically significant changes in vital sign - Pulse rate | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Beats per minute (BPM)
Incidence of clinically significant changes in vital sign - Body Temperature | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Celsius (°C)
Incidence of clinically significant changes in vital signs - Weight | Participants monitored throughout treatment period and during follow-up, up to 6 months
  Kilograms (kg)
Incidence of clinically significant changes in ECGs | Participants monitored throughout treatment period and during follow-up, up to 6 months
  QT interval (milli second (ms))

SECONDARY OUTCOMES:
Preliminary efficacy by means of RECIST evaluation | Participants monitored throughout treatment period every 6 weeks until disease progression, up to 6 months
  1. ORR will be assessed by monitoring tumor response and progression using RECIST v1.1
  2. ORR will be assessed by monitoring tumor response and progression using mRECIST
  3. ORR will be assessed by monitoring tumor response and progression using RECIST v 1.1 in liver lesions only
Plasma levels of α fetoprotein (AFP) | Participants monitored throughout treatment period every 6 weeks until disease progression, up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Plummer, Professor, Principal Investigator — Northern Institute for Cancer Research, Newcastle
Locations (18):
- Belgium (2):
  - Antwerp University Hospital, Antwerp
  - University Hospitals Gasthuisberg, Leuven
- South Korea (6):
  - CHA Bundang Medical Center, Gyeonggi-do
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (6):
  - Hospital Clinic Carrer Rosselló 161, Barcelona
  - Hospital Vall Hebrón, Barcelona
  - START Barcelona HM Nou Delfos, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid-FJD, Madrid
- United Kingdom (4):
  - Beatson West of Scotland Cancer Care, Glasgow
  - Guy's Hospital, Oncology and Clinical Trials, London
  - Northern Institute for Cancer Research, Newcastle upon Tyne
  - Chruchill Hospital, Cancer and Haematology Centre, Oxford

IPD SHARING:
Plan to Share IPD: Undecided